CLINICAL TRIAL: NCT01049932
Title: PrEP TMC278LA: Safety, Tolerability and Pharmacokinetics of TMC278LA in HIV Negative Volunteers
Brief Title: Pre-Exposure Prophylaxis Using TMC278LA
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial closed due to additional safety information.
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Marta Boffito, St Stephen's AIDS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSAT 037; EudraCT: 2009-017631-17 (Other: European Clinical Trials Database)
Record Dates: First submitted 2010-01-11; First posted 2010-01-15 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
Keywords: HIV; Human Immunodeficiency Virus (HIV); HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): TMC278LA 600mg injected intramuscularly (i/m)
  Interventions: Drug: TMC278LA

INTERVENTIONS:
Drug: TMC278LA — TMC278LA 600mg injected intramuscularly (i/m)
  Other Names: Rilpivirine

SUMMARY:
Pre-exposure prophylaxis (PrEP) is an experimental HIV-prevention strategy using antiretroviral (ARV) agents to protect HIV negative individuals from HIV infection.TMC278 is a new drug being developed for this type of HIV treatment. It is hoped that this drug may be used to help prevent HIV transmission in future. A 'long acting' formulation of TMC278 has been developed. Long acting means that the drug will be present in the blood for longer. It is this formulation of the drug that will be investigated in this study. Subjects will receive the drug by injection.

The purpose of this study is to investigate the safety of the drug and how well it is tolerated by the body. The study will look at the levels of the study drug in the subjects blood over the duration of the study.

DETAILED DESCRIPTION:
While for certain diseases, the use of medications by healthy people has been proven to function as prophylaxis, i.e. malaria, it is still unknown whether PrEP can help prevent HIV infection from exposure during sex or injection-drug use.

To address whether PrEP is safe and effective for use in humans, the traditional sequence of drug development steps should be followed as closely as possible.

TMC278 (rilpivirine) is a new investigational non nucleoside reverse transcriptase inhibitor (NNRTI) discovered and in development by Tibotec, a division of Johnson & Johnson. Data from clinical development (Phase IIB) suggest that TMC278 has a similar efficacy and better side-effect profile as compared to other, older, NNRTIs, such as efavirenz. Like TMC125 (etravirine), TMC278 is a diarylpyrimidine (DAPY - a class of molecule that resembles the pyrimidine nucleotides found in DNA, and which have shown potency in inhibiting the activity of HIV reverse transcriptase).

Tibotec is currently investigating TMC278 in two formulations: an oral formulation for HIV treatment and, in early phase, a long acting (LA) injectable formulation for HIV treatment. The latter has also potential application for HIV transmission prevention.

TMC278LA is an innovative drug formulation and its long apparent half life may allow administration of PrEP monthly rather than orally and daily, as for other ARV that are currently studied as PrEP agents.

Therefore, a phase I/II, open-label, prospective, single arm, pharmacokinetic clinical trial in 100 HIV negative subjects (50% of whom will have to be of self-identified African ancestry and 50% females, approximately) is to be conducted. The study will examine whether a monthly dose of TMC278LA not exceeding 600 mg i/m over a time period of approximately six months, with a loading regimen of the first two i/m injections separated by two weeks, is safe and well tolerated by HIV-negative subjects.

Investigation of drug pharmacokinetics in plasma and genital secretions will be also carried out in order to ensure optimal drug exposure during drug administration.

100 evaluable subjects will be enrolled, with approximately 50 of African ancestry, and 50 females. This will provide 50-subject-years of safety data in order to support a later large phase III global efficacy study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria within 42 days prior to the baseline visit:

1. Must understand and sign a written informed consent form, prior to participation in any screening procedures and must comply with all study requirements
2. Male or non-pregnant, non-lactating females of different ethnic backgrounds
3. Age between 18 to 50 years, inclusive
4. Body Mass Index (BMI) of 16 to 35 kg/m2, inclusive
5. Absence of any significant health problems on the basis of the screening procedures; including medical history, physical examination, vital signs, ECG
6. Clinically significant laboratory abnormalities
7. Willing to undergo HIV testing, HIV discussion and receive HIV test results (according to the "UK National Guidelines for HIV Testing 2008", www.bhiva.org)
8. Women of childbearing potential must be using an adequate method of contraception (diaphragm, intrauterine device, condoms, anatomical sterility in self or partner) to avoid pregnancy throughout the study and for a period of at least four months after the study follow up visit. Oral hormonal methods and implant contraceptives are allowed but only in combination with the additional protection of a barrier method
9. If sexually active male, willing to use an effective method of contraception such as condoms, anatomical sterility from the day of enrolment until at least four months after the follow up visit
10. Likely to remain resident in the UK for the duration of the study and follow-up period
11. Willing to consent to their personal details being entered onto The Over volunteering Prevention Scheme (TOPS) database
12. Willing to provide photographic identification at each visit.
13. Registered with a GP in the UK

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Any significant acute or chronic medical illness
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
3. Positive blood screen for syphilis, hepatitis A (IgM) B (HBs Ag) and/or C antibodies
4. Positive blood screen for HIV-1 and/or HIV-2 antibodies
5. High-risk behaviour for HIV infection which is defined as having one of the following within six months before study day 0 (first dose):

   i. had unprotected vaginal or anal sex with a known HIV infected person or a casual partner ii. engaged in sex work for money or drugs iii. acquired a sexually transmitted disease iv. having a high risk partner either currently or in the previous six months
6. Clinically relevant alcohol or drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events
7. Exposure to any investigational drug or placebo within 30 days of first dose of study drug (additional check to be made on TOPS www.tops.org.uk)
8. History of severe drug allergy that the Investigator thinks may increase the risk of developing an allergic reaction to the study drug
9. Use of any drug, including over-the-counter medications and herbal preparations, within two weeks prior to first dose of study drug unless approved by the Investigator
10. Females who are pregnant or lactating
11. Females of childbearing potential not using effective non-hormonal birth control methods, or not willing to practise these birth control methods for at least four months after the study follow up visit
12. Males unwilling to use an effective method of contraception such as condoms, anatomical sterility from the day of enrolment until at least four months after the follow up visit

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Local or systemic adverse events including local reactions to the IMP, all DAIDS (2004) grade ≥1 adverse events, serious adverse events (including laboratory abnormalities) and suspected unexpected serious adverse reactions (SUSARs) | 217 ± 10 days

SECONDARY OUTCOMES:
Drug plasma pharmacokinetics following first i/m dose and at steady state | 217 ± 10 days
Male and female genital tract drug concentrations following first i/m dose and at steady state | 217 ± 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust (London); Akil Jackson, Dr, Principal Investigator — St Stephen's AIDS Trust (London); Martin Fisher, Dr, Principal Investigator — Royal Sussex County Hospital, Brighton; Alan Winston, Dr, Principal Investigator — St Mary's Hospital, London; Julie Fox, Dr, Principal Investigator — St. Thomas's Hospital (London)
Locations (4):
- United Kingdom (4):
  - Royal Sussex County Hospital, Brighton, Sussex
  - St. Thomas's Hospital, London
  - St Stephen's Centre, London
  - St. Mary's Hospital, London